CLINICAL TRIAL: NCT03538639
Title: Vascular Disease Discovery Protocol
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 180108; 18-H-0108
Record Dates: First submitted 2018-05-25; First posted 2018-05-29 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12-05

CONDITIONS: Vascular Dysfunction; Genetic Mutations; Genetic Predisposition
Keywords: Etiology of Rare and Orphan Diseases with Vascular Phenotype; Natural History of Rare and Orphan Diseases with Vascular Phenotype; Pathophysiology of Uncommon Vascular Diseases; Undiagnosed Diseases; Rare Human Diseases with Vascular Features; Natural History
MeSH Terms: conditions — Genetic Predisposition to Disease; Undiagnosed Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: Adult index cases (affected) and relatives (affected and unaffected)
- 2: Child index cases (affected) and child relatives (affected and unaffected)
- 3: Healthy adult volunteers

SUMMARY:
Background:

Some genetic diseases put increase the risk of heart and blood diseases, which are the number one cause of death and disability in the U.S. Researchers want to study diseases of the heart and/or blood vessels. They want to collect data and specimens from affected people, their family members, and healthy people.

Objective:

To study diseases of the heart and/or blood vessels.

Eligibility:

People age 2 and older who may have genetic disease affecting the heart and/or blood vessels Their relatives

Healthy volunteers

Design:

Participants will be screened with a medical history, physical exams, and imaging tests. Participants may have a few visits or visits for 2 weeks or more. This will depend on their age and disease status. Visits may include:

Photographs of the face and body

Heart tests

Samples taken of blood, urine, saliva, skin, and/or tissue

Scans. For some, a dye may be injected into a vein.

A six-minute walk test

Lung tests. For some, participants will blow into a tube. For others, they will breathe in a gas from a mask, have a small injection, then have a scan.

Stress tests while walking on a treadmill or riding a stationary bike

Ultrasound of veins and arteries

Devices outside the body testing the stiffness and function of arteries

Eye exam and eye tests. For some, a dye may be injected in a vein.

Blood pressure tests

Measurements of blood flow under the skin and in the arms and fingernail blood vessels

Devices outside the body testing flexibility of the blood vessels and skin, and skin temperature

DETAILED DESCRIPTION:
The NIH provides a unique opportunity for research scientists to participate in the bench-to-bedside process, which is essential for the full implementation of translational medicine programs. The study of rare monogenetic and undiagnosed diseases is a complex bedside-to-bench-to-bedside endeavor. Recent studies show that rare genetic variants are more likely than common variants to have deleterious effects on protein structure, function, and/or expression, possibly leading to clinically relevant events. Studies of large patient populations offer the opportunity to identify rare genetic variants underlying human disease and will have impactful implications for human health. We propose to characterize the etiology and natural history of rare and orphan diseases with vascular phenotypes. We will also study rare genetic modifiers and identify novel disease mechanisms contributing to common vascular diseases. Subsequent disease-related protocols may be developed based on findings from subjects enrolled in this protocol for further intensive natural history studies and potential innovative therapeutic studies. In addition to its role in investigating individuals who are of interest to the Translational Vascular Medicine Branch (TVMB) of the NHLBI, this protocol can provide a possible avenue for admitting subjects from other NIH programs, such as the NIH Undiagnosed Diseases Program, the Center for Human Immunology Trans-institute program or other NIH protocols where subjects exhibit vascular phenotypes.

ELIGIBILITY:
* INCLUSION CRITERIA:
* All subjects must be between the ages of 2-100 years old.
* Affected pregnant women if they have been referred with a known or suspected pathology or if they become pregnant while on study.
* Unaffected related pregnant women (including spouses/partners) for cord blood and tissue collection (surgical waste) only at the time of delivery.

EXCLUSION CRITERIA:

* Healthy volunteers unable to give informed consent
* Healthy volunteers who decline to have blood drawn and/or tissue studies or who do not consent to have samples stored for future research.
* Cognitively impaired individuals who are not affected.
* Cognitively impaired individuals not related to affected subjects.

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We expect to enroll an unlimited number of subjects. The study population will be divided into groups that reflect both the potential studies that may be performed in distinct groups and the risk to benefit analysis for these groups. The appendices at the end of the protocol describe possible procedures and risk profiles for all the study subjects. Vulnerable populations, including pregnant women, children and cognitively impaired persons, may participate in this study. The groups include: 1.Adult index cases (affected) and relatives (affected and unaffected) 2.Child index cases (affected) and child relatives (affected and unaffected) 3.Healthy adult volunteers
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-07-30 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2037-05-15 (Estimated)

PRIMARY OUTCOMES:
Rapid initiation of new, disease-specific investigations to enable the collection of data and biospecimens on affected subjects, their family members and healthy controls, and to assist in the generation of diagnoses and further the understandin... | ongoing
  Understanding of disease pathophysiology in subjects with uncommon vascular disease presentation.

SECONDARY OUTCOMES:
to improve diagnosis, identify biomarkers, develop outcome measures, create centers of expertise and provide the foundation for therapy development. Clinically indicated procedures may yield data that can be used to support or guide research obj... | ongoing
  to improve diagnosis, identify biomarkers, develop outcome measures, create centers of expertise and provide the foundation for therapy development. Clinically indicated procedures may yield data that can be used to support or guide research objectives.

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Boehm, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2018-H-0108.html